CLINICAL TRIAL: NCT01482832
Title: Preventing Postpartum Depression in Adolescent Mothers
Brief Title: Interpersonal Therapy-Based Treatment to Prevent Postpartum Depression in Adolescent Mothers
Acronym: REACH 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Pacific Institute for Research and Evaluation (Other); Brown University (Other)
Responsible Party: Principal Investigator, maureen phipps, Study Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH093342 (NIH); R01MH093342 (NIH)
Record Dates: First submitted 2011-11-25; First posted 2011-12-01 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Postpartum Depression
Keywords: Randomized trial; Postpartum depression; Adolescent pregnancy; Interpersonal psychotherapy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Behavioral: Interpersonal therapy-based treatment Participants assigned to receive interpersonal therapy-based treatment will focus on the psychological aspects of pregnancy and factors that may play a role in the development of postpartum depression in teenage mothers, such as poor social support, role transitions, and life stressors. Both groups will attend 5 weekly sessions and have a brief booster session postpartum.
  Interventions: Behavioral: Interpersonal therapy-based treatment
- Control (Active Comparator): Behavioral: Standard care Participants assigned to receive standard care will focus on prenatal education including issues associated with pregnancy and postpartum. Both groups will attend 5 weekly sessions and have a brief booster session postpartum.
  Interventions: Behavioral: Interpersonal therapy-based treatment

INTERVENTIONS:
Behavioral: Interpersonal therapy-based treatment — Interpersonal therapy-based treatment Participants assigned to receive interpersonal therapy-based treatment will focus on the psychological aspects of pregnancy and factors that may play a role in the development of postpartum depression in teenage mothers, such as poor social support, role transitions, and life stressors. (5 weekly sessions with a booster session postpartum)
  Other Names: REACH 2

SUMMARY:
The Specific Aim of this study is to conduct a randomized controlled trial to evaluate whether Project REACH (an interpersonal psychotherapy-based intervention) compared with a didactic attention-control program reduces the risk of PPD in adolescent mothers.

Primary Hypothesis:

1. The intervention (Project REACH) will be significantly more efficacious than the control program in reducing the risk of PPD up to six months postpartum in adolescent mothers.

   Secondary Hypotheses:
2. The decreased rate of major depression in the Project REACH group compared to the control program group will be sustained through one year postpartum.
3. Adolescent mothers in Project REACH compared to the control program group will have higher levels of maternal-child bonding.

DETAILED DESCRIPTION:
Each year, more than 400,000 births in the United States are to mothers less than 20 years old. Alarmingly, approximately 25-36% of teen mothers experience postpartum depression (PPD), a condition associated with significant social and health morbidity. PPD places teen mothers and their children at great risk during an already challenging time in their lives. Preventing PPD in this vulnerable population is essential to improving overall health.

Project REACH is a randomized controlled trial, to evaluate whether our novel preventive intervention compared to a didactic attention control reduces the risk of PPD in adolescent mothers. The intervention, REACH (Relax, Encourage, Appreciate, Communicate, Help), is based on Interpersonal Psychotherapy (IPT) and targets those factors that may play a significant role in the development of PPD in adolescent mothers (i.e., poor social support, role transitions and life stressors). The control condition includes didactic prenatal education sessions.

Project REACH builds on the foundation of our NIMH-funded treatment development project and pilot study (R34 MH077588). The pilot study demonstrated feasibility, acceptability and initial efficacy in a small sample. The current R01 proposal aims to evaluate the efficacy of the Project REACH intervention in reducing the risk of PPD.

ELIGIBILITY:
Inclusion Criteria:

* Less than 24 weeks pregnant
* Not currently being treated for depression
* Speaks and reads English fluently

Exclusion Criteria:

* Currently receiving mental health services from a health care provider
* Meets DSM-IV criteria for an affective disorder, substance use disorder, or psychosis

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis of depression | within 6 months postpartum
  Outcome assessment using KID-SCID

SECONDARY OUTCOMES:
Degree of depressive symptoms | pre-randomization; 34-36 weeks gestation; within 4 days postdelivery; postpartum weeks 6, 12, 24 and 52
  Outcomes assessment using CDRS

CONTACTS AND LOCATIONS:
Overall Officials: Maureen G Phipps, MD, MPH, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Not at this point.

REFERENCES:
- [Derived] Phipps MG, Ware CF, Stout RL, Raker CA, Zlotnick C. Reducing the Risk for Postpartum Depression in Adolescent Mothers: A Randomized Controlled Trial. Obstet Gynecol. 2020 Sep;136(3):613-621. doi: 10.1097/AOG.0000000000004003. PMID 32769639